CLINICAL TRIAL: NCT00882219
Title: XERES Trial: Clinical Evaluation of Patients With Everolimus-eluting Stent " Xience V® " Implanted in the Treatment of Restenosis in Non-coated Metallic Stent (BMS In-stent Restenosis) During a 2 Year Clinical Follow-up Period
Brief Title: Clinical Evaluation of Patients With Everolimus-eluting Stent Xience V® Implanted in the Treatment of Restenosis in Non-coated Metallic Stent (BMS In-stent Restenosis) During a 2 Year Clinical Follow-up Period
Acronym: XERES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 330704
Record Dates: First submitted 2009-04-14; First posted 2009-04-16 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-09

CONDITIONS: Coronary Restenosis
Keywords: Drug eluting stent; Stents; Angioplasty; Chronic coronary occlusion; Stent thrombosis; Vascular disease; Myocardial ischemia; Coronary artery stenosis; Coronary Disease; Coronary Artery Disease; Coronary Restenosis
MeSH Terms: conditions — Coronary Restenosis; Vascular Diseases; Myocardial Ischemia; Coronary Stenosis; Coronary Disease; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Xience V® (Experimental)
  Interventions: Device: Xience V®

INTERVENTIONS:
Device: Xience V® — Placement of a Xience V® stent within a restenosed bare metal stent.

SUMMARY:
Interventional, prospective, non-randomized, non-comparative, open and multicentric study of patients with everolimus-eluting stent " Xience V® " implanted in the treatment of restenosis in non-coated metallic stent (BMS in-stent restenosis) during a 2 year clinical follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Patients affiliated to a social security or equivalent regimen
* Patients agreeing to participate in the study (Patient with signed informed consent )
* Patients with evidence of myocardial ischemia (stable or unstable angina, silent ischemia, positive functional exploration or a reversible modification in the ECG consistent with ischemia).
* Patient acceptable candidate for CABG surgery
* Patient agreeing to undergo all protocol scheduled follow-up examinations.
* Patients who tolerate the association Aspirin (dosed 75 to 160 mg/day) and Clopidogrel at 75 mg/day for at least 6 months

Angiographic inclusion criteria:

* Patient with de novo and sole in-stent restenosis (focal, diffuse or proliferative) in a non-coated metallic stent with or without any other coronary lesions.
* Patient with target reference vessel diameter between 2.5 and 4 mm by visual estimate
* Patient with a target lesion ≤ 22mm by visual estimate
* Patient with a target lesion in an artery with a visual estimate of the restenosis between 50 and 99% and a TIMI flow grade > 1
* Patient with multiple lesions, the other lesions have been treated with success

Exclusion Criteria:

* Patient in emergency
* Patient pregnant
* Patient nursing
* Patient unable to give informed consent personally.
* Patient with myocardial infarction within the previous 72 hours.
* Patient with limited life expectancy (lesser than 1 year post-inclusion)
* Patient with unstable arrhythmia
* Patient with left ventricular ejection fraction (LVEF) lesser than 30%
* Patient receiver of a cardiac or any other organ transplantation or candidate to an organ transplant
* Patient who receive or scheduled to receive chemo- or radio- therapy within the 30 days prior to any protocol-related procedure.
* Patient treated with immunosuppressives or for known immunodepressive or auto-immune pathologies
* Patient receiving chronically anticoagulant therapy with an INR greater than 2.5
* Patient with known hypersensitivity or contraindications to anti-platelet drugs, everolimus, heparin, chromium cobalt alloys, nickel, tungsten, acrylic- or fluoro- polymers or sensitivity to angiographic contrast agents.
* Patient with planned elective surgery requiring the interruption or discontinuation of anti-platelet therapy.
* Patient with platelet count <100 000/ mm3 or >700 000mm3 ; WBC counts <3 000/mm3 or known or suspected liver disease
* Patient with severe renal insufficiency (creatinine clearance rate < 30 ml/min), or under dialysis
* Patient with an history of coagulopathy refusing blood transfusion
* Patient who had a stroke/cerebrovascular accident or transient cerebrovascular ischemia in the preceding 6 months
* Patient with urinary or gastro-intestinal bleed in the preceding 6 months
* Patient with other known serious medical illness or known history of substance abuse (alcohol, drugs) that might result in non-compliance to the investigational plan, or interfere with the results or diminish the life expectancy to less than a year.
* Patient enrolled in an interventional study with another medical device or drug Angiographic exclusion criteria
* Patient with in-stent restenosis located on the left main on the coronary by-pass
* Patient with a lesion of the in-stent restenosis located in a bifurcation including a lateral branch of diameter > 1.5mm
* Patient with the target vessel totally occluded
* Patient with a lesion of the restenosis previously treated with another device (with the exception of balloon-tipped catheter) such as a cutting balloon, an atherectomy, laser, brachytherapy or any another medicated stent.
* Patient with thrombus in the target vessel
* Patient with aorto-ostiale lesions
* Patient with previous failures of multiple lesions treated by angioplasty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2009-03; Primary Completion 2011-03 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Evaluation by QCA (Quantitative Coronary Angiography) of in-stent late loss after the implantation of the stent XIENCE V® | 9 months

SECONDARY OUTCOMES:
Evaluation by IVUS (Intra Vascular Ultrasound) of the in-stent volume obstruction percentage (%VO) after the implantation of a XIENCE V® stent | 9 months
Evaluation by IVUS of the mean volume of neointimal hyperplasia after the implantation of a XIENCE V® stent | 9 months
Evaluation by QCA of the in-stent binary restenosis rate | 9 months
Evaluation of the in-segment binary restenosis rate | 9 months
Evaluation by QCA of in-segment late loss | 9 months
Evaluation by IVUS of the in-segment % volume obstruction after the implantation of the XIENCE V® stent | 9 months
Evaluation by IVUS of the rate of late incomplete apposition | 9 months
Document the number of confirmed stent thrombosis | 1, 8, 9, 12 and 24 months
-Document the number of confirmed revascularizations (TLR, TVR) | 1, 8, 9, 12 and 24 months
Document the rate of MACE | 1, 8, 9, 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Didier Carrie, MD, Principal Investigator — HOPITAL DE RANGUEIL - CHU
Locations (1):
- Hopital de Rangueil - Chu, Toulouse, France